CLINICAL TRIAL: NCT04549779
Title: Respiratory Sequelae and Analgesic Efficacy of Different Local Anesthetic Volumes in Ultrasound-guided Interscalene Brachial Plexus Block in Patients Presented for Shoulder Arthroscopy
Brief Title: Different Local Anesthetic Volumes in Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 34017/08/20
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Diaphragmatic Disorder
Keywords: Excursion; Diaphragm; Shoulder arthroscope; Postoperative analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The patients will be blinded to their groups.
  * An anesthesia resident who will not participate in the study and have no subsequent rule in it will help in the preparation of local anesthetic mixtures under strict aseptic precautions.
  * An assistant nurse who will be blinded to the study groups and will have no subsequent rule in it will help in the collection of the data of measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (low volume) (Experimental): patients will receive 5 ml levobupivacaine 0.25% in ultrasound-guided interscalene brachial plexus block
  Interventions: Procedure: Low volume interscalene brachial plexus block
- Group II (intermediate volume) (Experimental): patients will receive 10 ml levobupivacaine 0.25% in ultrasound-guided interscalene brachial plexus block
  Interventions: Procedure: Intermediate volume interscalene brachial plexus block
- Group III (high volume) (Experimental): patients will receive 15 ml levobupivacaine 0.25% ultrasound-guided interscalene brachial plexus block.
  Interventions: Procedure: High volume interscalene brachial plexus block

INTERVENTIONS:
Procedure: Low volume interscalene brachial plexus block — ultrasound-guided interscalene brachial plexus block with 5 ml levobupivacaine 0.25%
  Arms: Group I (low volume)
Procedure: Intermediate volume interscalene brachial plexus block — ultrasound-guided interscalene brachial plexus block with 10 ml levobupivacaine 0.25%
  Arms: Group II (intermediate volume)
Procedure: High volume interscalene brachial plexus block — ultrasound-guided interscalene brachial plexus block with 15 ml levobupivacaine 0.25%
  Arms: Group III (high volume)

SUMMARY:
This prospective randomized study will be carried out on 75 patients in our university hospitals presented for shoulder arthroscopy under general anesthesia and ultrasound-guided interscalene brachial plexus block.

All the patients will receive ultrasound-guided interscalene brachial plexus block with injection of local anesthetic volume according to the group of the patient

* Group I (25 patients): patients will receive 5 ml levobupivacaine 0.25% ISPB
* Group II (25 patients): patients will receive 10 ml levobupivacaine 0.25% ISPB
* Group III (25 patients): patients will receive 15 ml levobupivacaine 0.25% ISPB After ensuring adequate sensory and motor blockade, general anesthesia will be carried out.

The primary outcome measurement will be the incidence of diaphragmatic hemiparesis 30 minutes after performing the block detected by US assessment of diaphragmatic excursion and the secondary outcome will be the postoperative pain scores and opioid consumption.

DETAILED DESCRIPTION:
This prospective randomized double-blind study will be carried out on 75 patients who will be presented for shoulder arthroscopy in Tanta university hospitals over 9 months duration (September 2020- May 2021) which will be started immediately after obtaining the approval from the institutional Ethical Committee.

Informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

Patients will be randomly classified using a computer-generated software of randomization into 3 groups:

* Group I (25 patients): patients will receive 5 ml levobupivacaine 0.25% ISPB
* Group II (25 patients): patients will receive 10 ml levobupivacaine 0.25% ISPB
* Group III (25 patients): patients will receive 15 ml levobupivacaine 0.25% ISPB

Anesthetic technique The patients will be assessed preoperatively in the anesthesia clinic through history taking, examination, and appropriate investigation. Pulmonary function tests (PEFR, FEV1, FVC, and FEV1/FVC) will be performed preoperatively. On arrival of patients to the preparation room, an intravenous line will be established and a fluid preload will be started (7 ml/kg of lactated ringer solution) and the patient will be connected to monitor that consist of 5 leads ECG, non-invasive blood pressure, pulse oximeter, and temperature were applied.

The patients will lie supine with ultrasound assessment of the diaphragmatic excursion during quiet breathing, (excluding deep breathing, crying, participants with nasal obstruction, rhinorrhea, or cough, and participants with abdominal pain). Then midazolam 2 mg will be injected slow i.v with the application of nasal cannula (2-3 L/min) to the patient. Then, ultrasound-guided interscalene brachial plexus block will be done under aseptic precaution with an injection of the pre-prepared local anesthetic mixture with its volume according to the group of the patient.

The patients will be monitored for 30 minutes before induction of anesthesia, during which assessment of the sensory blockade will be carried out. The sensory block will be assessed by exposure to cold (ice piece) to the area of the shoulder and the upper arm. The motor block will be evaluated by determining patients ability to abduct the shoulder and flex the elbow against gravity (0 = no block Y full strength, 1 = partial block Y weak but able to abduct or flex against gravity, 2 = complete block Y no activity of muscle group). Preserved sensation to the cold or strength to abduct the shoulder after 30 minutes from performing the block at the area of the shoulder and upper arm will be considered as failed block and the patient will be excluded from the study. Ultrasound assessment of the diaphragmatic excursion during quiet breathing will be done again 30 minutes after performing the block.

Induction of anesthesia will be carried out after 3 minutes of pre-oxygenation through a well-fitted face mask using 80% oxygen by fentanyl 1 ug/kg, propofol 1.5 mg/kg, and atracurium 0.5 mg/kg to facilitate tracheal intubation. After securing the airway through a suitable sized endotracheal tube, the patient will be connected to a mechanical ventilator with its parameters adjusted to maintain the end-tidal carbon dioxide 34-38 mmHg. Maintenance of the anesthesia will be performed by isoflurane 1.2 % in a low flow gas mixture (1 L/min) composed of oxygen: air 1:1 and incremental doses of atracurium 0.1 mg/kg. A temperature probe will be inserted in the nasopharynx for core temperature monitoring. The depth of anesthesia will be monitored by the bispectral index (Covidien, Mansfield, MA, USA). The BIS values will be kept 40-60. An additional bolus dose of fentanyl 0.5 ug/kg was used in case of increase BIS more than 60 or increase in the heart rate or mean arterial pressure by more than 15 % of the baseline values.

At the end of the surgery, the isoflurane will be switched off with reversal of muscle relaxation by neostigmine 0.05 mg/kg and atropine 0.01 mg/kg with awake tracheal extubation and transfer of the patient to the recovery room for postoperative monitoring and supplementation of oxygen through nasal cannula (2-3 L/min). All the patients will receive 4 mg dexamethasone i.v after induction of anesthesia and 4 mg of ondansetron i.v at the end of the surgery to guard against postoperative nausea and vomiting. Also, paracetamol 1 gm i.v infusion every 6 hours will be given routinely to all patients in the postoperative period. In the PACU, ultrasound-guided assessment of the diaphragmatic excursion will be done. Also, pulmonary function (PEFR, FEV1, FVC, and FEV1/FVC) tests will be repeated before discharging the patients from the recovery room after exclusion of the effect of sedation by the aid of the modified observer¡¦s assessment of alertness.

Bradycardia (heart rate less than 50 b/min) will be managed by atropine 0.3 mg i.v) and hypotension (mean arterial pressure less than 65 mmHg or decrease by more than 20 % of the pre-anesthesia value) will be managed by ephedrine 10 mg i.v and i.v infusion of ringer lactate that may be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes aged (21-70 years) with ASA physical status I-III scheduled for shoulder surgeries.

Exclusion Criteria:

* Patients with COPD
* Sever bronchial asthma
* BMI > 40 kg/m2
* Mental dysfunction
* Allergy to local anesthetics
* Chronic opioid use
* Patients refusal

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
The incidence of diaphragmatic hemiparesis 3 | After 30 minutes of performing the block
  The incidence of diaphragmatic hemiparesis 30 minutes after performing the block detected by US assessment of diaphragmatic excursion

SECONDARY OUTCOMES:
The postoperative pain scores | Within the first 24 hours after surgery
  Postoperative Numerical rating score (NRS) every 2 hours in the first six hours, then every 4 h till 24 h. When NRS scores reach 4 or more, 3 mg of i.v tramadol will be given and can be repeated if required with calculation of the total postoperative morphine consumption in mg in the first 24 hours after surgery and the time to the first request of rescue analgesia.
The postoperative opioid consumption | Within 24 hours after surgery
  The total dose of tramadol consumed in the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Algharbia Governate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Access Criteria: Contact the principle investigator